CLINICAL TRIAL: NCT03626519
Title: Effects of Menthol on Dyspnoea Induced by Exercise in COPD Patients
Brief Title: Effects of Menthol on Dyspnoea in COPD Patients
Acronym: MEDiC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier du Havre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2018-A00585-50
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Copd; Dyspnea; Lung Diseases
Keywords: COPD; Menthol; Exercise; Dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Lung Diseases; Motor Activity | interventions — Menthol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test with Menthol (Experimental): Patients will chew a menthol flavored chewing gum 5 minutes before perform one Six-minute Walk Test
  Interventions: Other: Test with Menthol
- Test with placebo (Placebo Comparator): Patients will chew a strawberry flavored chewing gum 5 minutes before perform one Six-minute Walk Test
  Interventions: Other: Test with placebo

INTERVENTIONS:
Other: Test with Menthol — patients will perform a Six-minute walk test according to American Thoracic Society guidelines
  Arms: Test with Menthol
Other: Test with placebo — patients will perform a Six-minute walk test according to American Thoracic Society guidelines
  Arms: Test with placebo

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is characterised by non-reversible bronchial obstruction associated with systemic disorders and comorbid factors. Dyspnoea is a common symptom among patients with Chronic Obstructive pulmonary Disease (COPD). Dyspnea is the primary symptom limiting exercise and daily activities in these patients. It has been reported that breathing cold air could decrease dyspnoea induced by exercise and could improve exercise performance. The aim of this study is to carry out the effect of cooling sensation induced by menthol chewing-gum on dyspnoea and exercise performance among patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of COPD
* Dyspnea in daily living (2-4 on the modified medical research council dyspnea scale)
* Clinically stable

Exclusion Criteria:

* exercise contraindication Any musculoskeletal problems, cardiovascular or neurological comorbidities that limits exercise.
* exacerbation during the study
* Inability to chew or patients with swallowing disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Change in Dyspnea after each tests | The outcome will be measured before and at the end of the test, the two six-minute walk test will perform the same day, separate from 30 minutes minimum for a total time frame of 1 day.
  Change in dyspnea using Modified Borg Scale (0 - 10 points) 0=no dyspnea ; 10 = maximal effort

SECONDARY OUTCOMES:
Change in respiratory rate | Data will be continuously collected during every tests. The two six-minute walk test will perform the same day, separate from 30 minutes minimum for a total time frame of 1 day.
  Change in respiratory rate (cycles per minute) will be measured breath-by-breath using a Respiratory Inductive Plethysmography
Change in inspiratory capacity | The outcome will be measured before and at the end of the test, the two six-minute walk test will perform the same day, separate from 30 minutes minimum for a total time frame of 1 day.
  Change in inspiratory capacity (Liters) will be measured using a portable spirometer
Change in Cardiac Frequency | Data will be continuously collected during every tests. The two six-minute walk test will perform the same day, separate from 30 minutes minimum for a total time frame of 1 day.
  Change in Cardiac Frequence (bpm) using a pulse oximetry
Change in Oxygen Saturation | Data will be continuously collected during every tests. The two six-minute walk test will perform the same day, separate from 30 minutes minimum for a total time frame of 1 day.
  Change in Oxygen Saturation (%) using a pulse oximetry
Change in tidal volume | The outcome will be measured before and at the end of the test, the two six-minute walk test will perform the same day, separate from 30 minutes minimum for a total time frame of 1 day.
  Change in tidal volume (Liters) will be measured breath-by-breath using a portable spirometer
Change in 6-min walk distance | The outcome will be measured at the end of each tests. The two six-minute walk test will perform the same day, separate from 30 minutes minimum for a total time frame of 1 day.
  Change in 6-min walk distance (meters).

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Prieur, Principal Investigator — Groupe Hospitalier du Havre; Marc Beaumont, Principal Investigator — Centre Hospitalier des Pays de Morlaix; Mathieu Delorme, Principal Investigator — Resp'Air, Talence
Locations (3):
- France (3):
  - Centre hospitalier des Pays de Morlaix, Morlaix, Brittany Region
  - Groupe Hospitalier du Havre, Le Havre, Normandy
  - Resp'Air, Talence, Nouvelle-Aquitaine

IPD SHARING:
Plan to Share IPD: Yes
Data type : deidentified participtant data
Supporting Information: CSR
Time Frame: after publication
Access Criteria: the request shall be sent to Guillaume Prieur (gprieur.kine@gmail.com)